CLINICAL TRIAL: NCT02328014
Title: A Phase 1/2 Proof-of-Concept Study of the Combination of ACP-196 and ACP-319 in Subjects With B-cell Malignancies
Brief Title: Acalabrutinib (ACP-196) in Combination With ACP-319, for Treatment of B-Cell Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-001
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Non-Hodgkins Lymphoma; Multiple Myeloma; B-All
Keywords: Bruton tyrosine kinase inhibitor; Btk; B-Cell Malignancies; Mantle Cell; Multiple Myeloma; CLL; SLL; DLBCL; Follicular; Waldenstrom; B-All
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — acalabrutinib; N-(1-(7-fluoro-2-(pyridin-2-yl)quinolin-3-yl)ethyl)-9H-purin-6-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): The acalabrutinib dose will be fixed and the ACP-319 dose will be escalated in each of three cohorts, and each cohort will take both study drugs by mouth, twice per day (BID) at approximately 12 hour intervals.
  Expansion groups of up to 12 subjects for Germinal center B-cell (GCB) DLBCL and Non-GCB DLBCL to take a fixed dose of acalabrutinib and ACP-319. Each disease group will take both study drugs by mouth, twice per day (BID) at approximately 12 hour intervals.
  Interventions: Drug: Acalabrutinib; Drug: ACP-319

INTERVENTIONS:
Drug: Acalabrutinib — Oral
  Other Names: ACP-196
Drug: ACP-319 — Oral

SUMMARY:
This study is evaluating the safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy acalabrutinib and ACP 319 in B-cell malignancies.

DETAILED DESCRIPTION:
Part 1, Dose Escalation, is comprised of 3 dosing cohorts of 6 subjects each. Acalabrutinib dosing is fixed in all cohorts at 100 mg PO twice daily (BID). In addition to acalabrutinib, subjects in Cohort 1 will receive ACP-319, 25 mg BID; Cohort 2 will receive ACP-319, 50 mg BID: and Cohort 3 will receive ACP-319 100 mg BID. The maximum tolerated dose (MTD) of the study treatment combination will be determined by assessing dose-related toxicities (DLTs) for each cohort at the end of Cycle 1 prior to dose escalation. If there are greater than or equal to 2 DLTs in a cohort, dose escalation will not occur and the MTD will be the highest daily dose for which less than 33% of the subjects in that cohort experienced DLTs in Cycle 1.

Part 2, Dose Expansion, includes 12 subjects per histology, dosing at the MTD for the combination of acalabrutinib and ACP-319 established in Part 1. Subjects will continue dosing until disease progression or unacceptable drug-related toxicity.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of a b-cell malignancy as documented by medical records and with histology based on criteria established by the World Health Organization (WHO).
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use contraception during the study and for 90 days after the last dose of study drugs if sexually active and able to bear or beget children.

Exclusion Criteria

* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of study drugs, or put the study outcomes at undue risk.
* Central nervous system (CNS) involvement by lymphoma/leukemia
* Any therapeutic antibody within 4 weeks of first dose of study drugs.
* The time from the last dose of the most recent chemotherapy or experimental therapy to the first dose of study drugs is < 5 times the half-life of the previously administered agent(s).
* ANC < 0.5 x 10^9/L or platelet count < 50 x 10^9/L unless due to disease involvement in the bone marrow.
* Creatinine > 1.5 x institutional upper limit of normal (ULN); total bilirubin > 1.5 x ULN (unless due to Gilbert's disease); and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3.0 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2025-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Clinical Study Infromation Center, Study Director — 1-877-240-9479 - information.center@astrazeneca.com
Locations (7):
- United States (7):
  - Research Site, Orange, California
  - Research Site, Bethesda, Maryland
  - Research Site, Rochester, New York
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-001&attachmentIdentifier=24973127-5a2c-4c38-b322-8d5862f379df&fileName=ACE-LY-001_SAP-v1_Redacted.pdf&versionIdentifier=
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-001&attachmentIdentifier=903010aa-8039-41ba-9be1-5375d02fa590&fileName=ACE-LY-001-CSR-Synopsis_Redacted.pdf&versionIdentifier=
- See also: redacted study protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-001&attachmentIdentifier=00a8f454-eb32-4da4-9d56-70d3a689b3a2&fileName=ACE-LY-001_CSP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All data collection and Final analysis for the study has been completed. However, as we face a unique challenge in oncology studies, some patients benefiting from the medication, continue to receive treatment beyond final analysis with NO requirement for any further data collection or additional data analysis.
Groups:
- Part 1 Cohort 1: Part 1 Cohort 1: ACP-196 100 mg BID + ACP-319 25 mg BID continuously
- Part 1 Cohort 2: Part 1 Cohort 2: ACP-196 100 mg BID + ACP-319 50 mg BID continuously
- Part 1 Cohort 3: Part 1 Cohort 3: ACP-196 100 mg BID + ACP-319 100 mg BID continuously
- Part 2: Part 2: ACP-196 100 mg BID + ACP-319 50 mg BID continuously
Period: Overall Study
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2
Started | 6 | 6 | 6 | 22
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 22
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Disease Progression | 1 | 0 | 1 | 3
Not completed — Study Terminated by Sponsor | 4 | 1 | 1 | 0
Not completed — Subject Started Another Cancer Therapy | 0 | 5 | 4 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated = subjects who receive at least 1 dose of study drug; Efficacy evaluable = all-treated population with one evaluable response assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (7.3) | 68.0 (9.9) | 62.5 (7.9) | 68.3 (9.2) | 68.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 9 | 16
  Male | 3 | 5 | 3 | 13 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 6 | 22 | 39
  Not Reported | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 6 | 5 | 5 | 18 | 34
  Not Reported | 0 | 1 | 1 | 3 | 5
Region of Enrollment [Number; unit: Participants]
  United States | 6 | 6 | 6 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Best Response and Overall Response Rate
Description: Best response and overall response rate per the criteria investigator uses for each disease histology. Standardized response and progression criteria is based on established criteria for B-cell malignancies, including WM (Cheson 2014; Owen 2013; Hallek 2008; Bladé 1998; and Durie 2006).
Time Frame: from the start of the treatment to the last evaluable disease assessment, an average of 1 year
Population: All-Treated Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 22
percentage of participants
  CR | 33.3 [4.30 to 77.7] | 0 [0 to 45.9] | 16.7 [0.4 to 64.1] | 18.2 [5.2 to 40.3]
  VGPR | 16.7 [0.4 to 64.1] | 0 [0 to 45.9] | 0 [0 to 45.9] | 0 [0 to 15.4]
  PR | 33.3 [4.3 to 77.7] | 50 [11.8 to 88.2] | 50 [11.8 to 88.2] | 22.7 [7.8 to 45.4]
  SD | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 0 [0 to 45.9] | 4.5 [0.1 to 22.8]
  PD | 0 [0 to 45.9] | 33.3 [4.3 to 77.7] | 0 [0 to 45.9] | 36.4 [17.2 to 59.3]
  Missing | 0 [0 to 45.9] | 0 [0 to 45.9] | 33.3 [4.3 to 77.7] | 0 [0 to 15.4]
  ORR (CR+VGPR+PR) | 83.3 [35.9 to 99.3] | 50 [11.8 to 88.2] | 66.7 [22.3 to 95.7] | 40.9 [20.7 to 63.7]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days post last dose, an average of 1 year
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 4/22
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 5/6 | 11/22
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1 (N=6) | Part 1 Cohort 2 (N=6) | Part 1 Cohort 3 (N=6) | Part 2 (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary nocardiosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1 (N=6) | Part 1 Cohort 2 (N=6) | Part 1 Cohort 3 (N=6) | Part 2 (N=22)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (9)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 1 (1) | 2 (2) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (3)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 4 (5) | 4 (8) | 12 (20)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 2 (2) | 4 (5) | 5 (7)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0) | 8 (9)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 2 (3) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 2 (2) | 4 (7)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal disease carrier (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (4)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary nocardiosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (8) | 1 (1) | 4 (9) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 2 (3)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 4 (7) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (9) | 2 (6) | 12 (20)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (9) | 2 (5) | 10 (14)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure orthostatic decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (4) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6) | 2 (2) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 3 (4) | 6 (8)
Hemiapraxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (6) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 9 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT02328014/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT02328014/SAP_001.pdf